CLINICAL TRIAL: NCT02026726
Title: Oral Steroid Dose Pack Used As A Predictor For The Effectiveness Of Epidural Steroid Injections
Brief Title: Do Oral Steroid Dose Packs Predict How Well Epidural Steroid Injections Will Work?
Status: Terminated | Type: Observational
Why Stopped: could not recruit
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Bert L. Fichman, Staff Physician, Dartmouth-Hitchcock Medical Center
Other Study IDs: D11158
Record Dates: First submitted 2013-12-30; First posted 2014-01-03 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Lumbar Spine Disc Herniation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to show whether a standard oral steroid dose pack can be used as a screening tool to assess the effectiveness of a subsequent epidural steroid injection (ESI). If an oral steroid does not give a patient significant temporary relief of pain from a herniated lumbar disc then an epidural steroid injection will not either. Therefore the risk and expense associated from the interventional pain management procedure for those patients could be avoided and other treatment modalities pursued.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosed by participating physicians during the study enrollment period as having intervertebral disk herniation and persistent symptoms with or without some nonoperative treatment for at least 4 weeks
* Radicular pain (below the knee for lower lumbar herniations, into the anterior thigh for upper lumbar herniations)
* Evidence of nerve-root irritation with a positive nerve-root tension sign (straight leg raise-positive between 30° and 70°) or a corresponding neurologic deficit (asymmetrical depressed reflex, decreased sensation in a dermatomal distribution)
* Undergone either MRI or CT scan showing disc herniation (protrusion, extrusion, or sequestered fragment) at a level and side corresponding to the clinical symptoms
* Patients with multiple herniations can be included if only one of the herniations is considered symptomatic
* Preenrollment nonprocedural care can include: education/counseling, physical therapy, chiropractic therapy, anti-inflammatory medications, opioid analgesics, adjuvant analgesics such as anticonvulsants and antidepressants

Exclusion Criteria:

* Prior lumbar surgery
* Cauda equina syndrome
* Vertebral fractures
* Spine infection or tumor
* Severe motor deficit
* Inflammatory spondyloarthropathy
* Pregnancy
* Cardiac or pulmonary comorbid conditions contraindicating interventional procedures
* Diabetes
* Inability/unwillingness to have spinal injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that had magnetic resonance imaging (MRI) documented lumbar herniated discs with unilateral radicular symptoms that correlated to their physical exam and MRI findings.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Pain | Baseline,1 wk post oral steroid completion, 2 wks post ESI #1, 2 wks post ESI #2, 2 wks post ESI #3, then at 6 wks, 12 wks, 6 mo. & 12 mo. after last transforaminal ESI (TRESI).
  The primary endpoint will be a patient-reported pain as measured by a 10 cm visual analog scale (VAS) with 0 being no pain and 10 being the most severe pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Bert L. Fichman, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States